CLINICAL TRIAL: NCT07030205
Title: Resting-state Imaging and OSteoporosiS
Acronym: ROSS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RBHP 2025 PICKERING_ME; 2025-A00106-43 (Other: 2025-A00106-43)
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Resting state fMRI (rs-fMRI); Cognition
MeSH Terms: conditions — Osteoporosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Patient will have two visits :
  Visit 1 - Inclusion visit (informed consent, medical examination, stool sample and test/questionnaires assessing cognition, pain, physical activity, sleep, quality of life, anxiety and depression).
  -Visit 2 - End of study visit During this visit, a resting-State Functional Magnetic Resonance Imaging will be conducted.
  Postmenopausal healthy volunteers will have three visits :
  Visit 1 - Inclusion visit (informed consent, medical examination and bone density test) Visit 2 : stool sample and test/questionnaires assessing cognition, pain, physical activity, sleep, quality of life, anxiety and depression)
  -Visit 3 - End of study visit During this visit, a resting-State Functional Magnetic Resonance Imaging will be conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Postmenopausal Healthy volunteers (Experimental): 22 postmenopausal healthy women, matched by age, menopausal status, socio-educational level and manual laterality, will be included in this study
  Interventions: Other: Blood sample; Other: Bone density exam; Other: Tests and questionnaires of study; Other: Functional connectivity value of brain networks at rest
- Postmenopausal osteoporotic patients with fracture (Experimental): 22 Postmenopausal osteoporosis patients with fractures will be included in this study
  Interventions: Other: Blood sample; Other: Tests and questionnaires of study; Other: Functional connectivity value of brain networks at rest
- Postmenopausal osteoporotic patient without fracture (Experimental): 22 Postmenopausal osteoporosis patients without fractures will be included in this study.
  Interventions: Other: Blood sample; Other: Tests and questionnaires of study; Other: Functional connectivity value of brain networks at rest

INTERVENTIONS:
Other: Blood sample — A blood sample (fasting), for biobanking purposes to measure certain bone biological markers known to be indicators of bone remodeling (osteocalcin, sclerostin, periostin, irisin, procollagen type 1 N-terminal propeptide (P1NP), Dickkopf-related protein 1 (DKK1), and collagen type 1 C-terminal telopeptides (CTX)).
Other: Bone density exam — A bone density exam will be performed in order to verify the non-osteoporotic status of the healthy volunteers group.
  Arms: Postmenopausal Healthy volunteers
Other: Tests and questionnaires of study — An assessment of cognitive functions will be realized using Montreal Cognitive Assessment (MoCA), Cantab® tests (MOT, MTS, RTI, DGS), the Trail Making Test (TMT), verbal fluency, the Stroop test, the Dubois 5-word test, and the oral picture naming test. Other questionnaires will be used, assessing: sleep quality (Pittsburgh Physical Activity Questionnaire (PSQI)), anxiety and depression (the anxiety/depression scale (HAD)), quality of life (Short Form-36 quality of life questionnaire (SF-36)), physical activity (International Physical Activity Questionnaire (IPAQ)), and pain with the Brief Pain Inventory questionnaire (BPI) and the numerical scale (EN).
Other: Functional connectivity value of brain networks at rest — A Resting-State Functional Magnetic Resonance Imaging will be conducted in order to evaluate and compared functional connectivity value of brain networks at rest between three groups.

SUMMARY:
This study will be conducted in 20 postmenopausal healthy volunteers, 20 postmenopausal osteoporotic patients with fracture and 20 postmenopausal osteoporotic women without fracture, in order to compare functional connectivity between brain areas. Participants will complete different questionnaires and tests assessing cognition, quality of life, sleep, physical activity, pain, anxiety and depression. A biological sample will be performed in order to evaluate different markers of bone remodeling. A Resting-state functional magnetic resonance imaging (rs-fMRI) will be realized in order to establish functional connectivity between brain regions.

ELIGIBILITY:
Inclusion Criteria (patients):

* Women aged 50 or over, with postmenopausal osteoporosis, fractured or not, diagnosed by their rheumatologist,
* Able to give informed consent to participate in the research,
* Affiliation with the French Social Security.

Inclusion Criteria (healthy volunteers):

* Women aged 50 or over,
* Bone densitometry performed as part of the protocol, not suggestive of osteoporosis and validated by investigators,
* Matched to patients by age, menopausal status, socio-educational level and manual laterality,
* Able to give informed consent to participate in the research,
* Affiliation with the French Social Security.
* Registration or acceptance of registration in the national register of volunteers participating in Research.

Exclusion Criteria (patient and healthy volunteers):

* Presence of pacemaker,
* Presence of medical devices (implants or prostheses),
* Incompatibility of the patient with the safety criteria of the medical imaging center for carrying out magnetic resonance experiments at 3 Tesla,
* Contraindications to the realization of MRI without injection such as claustrophobia proven, hearing aid, pacemaker wearers, wearing a brain clip,
* Refusal to be informed in the event of the accidental discovery of an anomaly during the resting state functional magnetic resonance imaging,
* Woman under legal protection or deprived of liberty,
* Refusal to participation

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Functional connectivity value of brain networks at rest | At visit 2 (end of study visit, up to fifteen days after inclusion) for osteoporotic patient group and at visit 3 (end of study visit, up to one month after inclusion) for healthy volunteers group.
  The primary outcome is the functional connectivity value of brain networks at rest, calculated from resting-state fMRI data.

SECONDARY OUTCOMES:
Evaluation of cognitive function (MoCA test) | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  The Montreal Cognitive Assessment (MoCA) is the most sensitive rapid assessment test, with the broadest range of cognitive functions (attention, concentration, executive functions, memory, language, visuo-constructive abilities, abstraction, calculation, orientation). Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points; a score of 26 or above is considered normal.
Evaluation of cognitive function (Cantab test: MOT) | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  The Motor Screening Task provides a general assessment of whether sensorimotor deficits or lack of comprehension, will limit the collection of valid data from the participant. Coloured crosses are presented in different locations on the screen, one at a time. The participant must select the cross on the screen as quickly and accurately as possible. Outcome measures cover accuracy (Euclidean distance between finger and target) and difficulty speed adjustment.
Evaluation of cognitive function (CANTAB test: Reaction Time (RTI) | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  Reaction Time provides assessments of motor and mental response speeds, as well as measures of movement time, reaction time, response accuracy and impulsivity. The participant must select and hold a button at the bottom of the screen. Circles are presented above (one for the simple mode, and five for the five-choice mode). In each case, a yellow dot will appear in one of the circles, and the participant must react as soon as possible, releasing the button at the bottom of the screen, and selecting the circle in which the dot appeared. Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants.
Evaluation of cognitive function (CANTAB test: Digit Span) | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  Digit Span (DGS) is a measure of verbal short term and working memory. The participant will hear a sequence of digits and then immediately be prompted to verbally repeat the sequence, either as it was heard (forwards), or in reverse order (backwards). If the participant responds correctly, the next trial presents a longer sequence. The task terminates when participants responded incorrectly on three occasions at a span length. The participant's span is the longest number of sequential digits that can accurately be remembered. Outcome measures include the direction of the task (forwards or backwards), the longest sequence successfully reached and passed, and the total number of attempts.
Evaluation of cognitive function (CANTAB test: Match to Sample Visual Search) | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  Match to Sample Visual Search assesses attention and visual searching, with a speed accuracy trade-off. The participant is shown a complex visual pattern in the middle of the screen. After a brief delay, a varying number of similar patterns are shown in a circle of boxes around the edge of the screen. Only one of these patterns matches the pattern in the centre of the screen, and the participant must indicate which it is by selecting it. The outcome measures for this task cover accuracy and reaction time.
Evaluation of cognitive function (Trail Making Test) | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  The Trail Making Test is a neuropsychological test of visual attention and task switching. It can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning. There are 2 parts to the TMT. Both parts of the Trail Making Test consist of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1-13) and letters (A-L); The subject must correctly connect the circles as quickly as possible, within a limit of 100 seconds for part A and 300 seconds for part B. For each part, the completion time and the number of errors are collected.
Evaluation of cognitive function (Stroop test) | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  The Stroop Color Test assesses selective attention and the ability to inhibit cognitive interference, which occurs when the processing of one feature of a stimulus affects the simultaneous processing of another feature of the same stimulus. This test consists of three conditions:
  1. Color Naming (the instruction is to name the color of green, red, and blue squares),
  2. Reading "color name" words (the words "red," "blue," and "green" are printed in black),
  3. Interference (the instruction is to name the ink color of the "color name" words, printed in a different ink color-for example, the word "blue" is printed in red).
  For each condition, a sheet of 50 items is presented to the participant, and the total time is recorded (within a limit of 90 seconds for Conditions 1 and 2, and 180 seconds for Condition 3), as well as the number of corrected and uncorrected errors.
Evaluation of cognitive function (Verbal fluency test) | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  Verbal fluency is used to assess executive functions. This test is a simple language production test. This test assesses semantic fluency or categorical fluency. This is done by asking the participant to name as many nouns as possible in a given category in two minutes. Words from the same family and proper nouns should not be mentioned, and the participant should not repeat themselves. A score will be calculated based on the number of words given and the number of errors made.
Evaluation of cognitive function (5 words test) | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  The 5-word test is divided into two different stages. The first allows us to check the encoding of the information to be remembered. To do this, the subject will be shown a list of 5 words that they will have to read aloud and remember. To ensure memorization, the subject will be immediately questioned about the words they have just remembered. If necessary, clues may be provided. Once this first stage is completed, an intercurrent attentional test will be carried out. Its purpose is to divert the subject's attention for a sufficient time (between 3 and 5 minutes). At the end of the intercurrent test, the participant is again asked for the 5 words they previously remembered. Once again, clues may be provided if necessary. The data collected are the scores for immediate recall and delayed recall, with and without cueing.
Evaluation of cognitive function (Oral Picture Naming Test) | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  The oral picture naming test highlights the extent of the patient's potential word deficit and provides valuable insights into the process of impaired speech when analyzing the nature of the errors. During this test, the subject will be presented with cards representing objects. The subject must name the object presented. In this study, 20 cards will be presented to the participants. The data collected include the number of correctly named images and the type of errors.
The Pittsburgh Sleep Quality Index (PSQI) | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  The PSQI is a self-administered questionnaire with 19 items. It was developed to measure sleep quality in the month prior to the patient interview. This questionnaire includes 7 components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, hypnotic medication use and daytime dysfunction.
  The global score (0 to 21) is obtained by adding the sub-scores of the 7 components, each ranging from 0 to 3 points. In the absence of an answer to one or more questions, the subtotal using this question cannot be calculated and will affect the overall score.
  The higher the overall score, the greater the impairment in sleep quality. An overall score >5 is an indicator of sleep disturbance.
Evaluation of pain: The Brief Pain Inventory Questionnaire (BPI) | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  This self-assessment scale allows the patient to characterize the pain in terms of its intensity and its psychosocial repercussions by means of 11 scales rated from 0 (no pain or does not bother) to 10 (the most horrible pain you can imagine or completely bothers you).
  The BPI also asks the patient to black out the painful areas on a diagram (front and back) and to put an "S" if the pain is on the surface or a "P" if it is deep. The questionnaire also asks the patient to indicate what treatment or medication he or she is taking for the pain and what percentage improvement has been obtained.
Evaluation of pain: Numerical pain scale | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  This scale allows the patient to rate the pain on a scale with a minimum score of 0 (no pain) and a maximum score of 10 (worst pain).
Evaluation of quality of life: The 36-Item Short Form Survey (SF-36) | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  The quality of life of patients is assessed by the general questionnaire 36-Item Short Form Survey (SF-36) which can be administered by self or hetero-questionnaire. The SF-36 questionnaire was developed from the Medical Outcome Study, a 149-item questionnaire that was developed to assess how the American healthcare system affects the outcome of care. The SF-36 questionnaire is composed of 36 items and makes it possible to assess the physical and mental health of an individual using eleven questions relating to eight aspects of health: Physical activity, limitations due to physical state, physical pain, perceived health, vitality, life and relationship with others, limitations due to the mental state and mental health. Scores between 0 and 100 are determined. Scores tending towards 100 indicate a better quality of life.
Evaluation of anxiety and depression: The Hospital Anxiety and Depression Scale (HAD) | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  It is a self-administered questionnaire completed by the patient and based on the Hamilton scale. The HAD scale is a tool for screening for anxiety and depressive disorders. It includes 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus making it possible to obtain two scores (maximum score for each score = 21).
  To screen for anxiety and depressive symptomatology, the following interpretation can be proposed for each of the scores (A and D): ≤ 7: normal case; 8 to 10: borderline case; ≥ 11: abnormal case.
Evaluation of physical activity: International Physical Activity Questionnaire - Short Form | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  IPAQ assesses physical activity undertaken across a comprehensive set of domains including leisure time, domestic and gardening (yard) activities, work-related and transport-related activity; The IPAQ short form asks about three specific types of activity undertaken in the three domains introduced above and sitting. The specific types of activity that are assessed are walking, moderate-intensity activities and vigorous intensity activities; frequency (measured in days per week) and duration (time per day) are collected separately for each specific type of activity. The items were structured to provide separate scores on walking; moderate-intensity; and vigorous-intensity activity as well as a combined total score to describe overall level of activity. Computation of the total score requires summation of the duration (in minutes) and frequency (days) of walking, moderate-intensity and vigorous-intensity activity.
Sclerostin dosage | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  The dosage of sclerostin (pg/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes.
Osteocalcin dosage | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  The dosage of osteocalcin (µg/L) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 6 mL EDTA tube.
Periostin dosage | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  The dosage of periostin (pg/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes.
Irisin dosage | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  The dosage of irisin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken on 4 mL heparin tube for irisin dosage.
N-terminal propeptide of procollagen type 1 dosage | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  The dosage of N-terminal propeptide of procollagen type 1 (P1NP) (µg/l) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Dickkopf-related protein 1 dosage | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  The dosage of Dickkopf-related protein 1 (pg/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
C-terminal telopeptides of collagen type 1 dosage | At inclusion visit (Day 0) for osteoporotic patient group and at visit 2 (up to fifteen days after inclusion) for healthy volunteers group.
  The dosage of C-terminal telopeptides of collagen type 1 (CTX) (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 6 mL EDTA tube.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Eva Pickering, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No